Statistical Analysis Plan

Study Name:

Urgent Care Management of Respiratory Illness Enabled with Novel Testing Pathway

(URGENT): A Randomized Control Trial of Respiratory PCR versus Standard Care

**Date:** 13-Feb-2024

NCR: NCR213901

**Principal Investigator:** 

Name: Andrew C. Meltzer MD, MS

Title: **Associate Professor of Emergency Medicine** 

**George Washington University** Institution:

Statistical analysis: Categorical variables are expressed as absolute frequencies and

percentages. Continuous variables are presented as the mean and standard deviation

(SD) or as the median and interquartile range (IQR) when not normally distributed.

Categorical variables were compared using the chi-squared test or Fisher's exact test.

Continuous variables were compared using the Student's *t*-test or Mann–Whitney U

test, according to the Kolmogorov–Smirnov test of normality. All results were considered

statistically significant at P < 0.05. All analyses were performed using R version 4.1.1

(Comprehensive R Archive Network). The sample size was based on the expected high

satisfaction for time to result in 90% of patients in the syndromic assessment group

versus 60% of those in the SOC group with a power of 0.8 and a significance value of

0.05.